CLINICAL TRIAL: NCT06974526
Title: Randomized, Multicenter, Double-blind, Parallel, Placebo-controlled Study to Investigate the Safety and Exploratory Efficacy of the Absorbable Oxandrolone Implant as an Adjuvant Treatment in Rehabilitation Following Anterior Cruciate Ligament (ACL) Surgical Reconstruction (IMOX Study)
Brief Title: Subdermal Implant-bioabsorbable Oxandrolone Pellet For Rehabilitation Following Anterior Cruciate Ligament (ACL) Surgical Reconstruction
Acronym: IMOX
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Science Valley Research Institute (Other)
Collaborators: Stin Pharma (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IMOX
Record Dates: First submitted 2025-04-28; First posted 2025-05-16 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Anterior Cruciate Ligament (ACL) Reconstruction
Keywords: Anterior cruciate ligament (ACL); Oxandrolone; Absorbable subdermal implant; Adverse effects
MeSH Terms: interventions — Oxandrolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oxandrolone (Experimental): Absorbable oxandrolone implant (subdermal insertion) Men: 400 mg oxandrolone (two 200 mg oxandrolone implants each) Women: 200 mg oxandrolone (one 200 mg oxandrolone implant)
  Interventions: Drug: Oxandrolone
- Placebo (Placebo Comparator): Absorbable placebo implant (excipients; subdermal insertion) Men: 400 mg placebo (two 200 mg placebo implants each) Women: 200 mg placebo (one 200 mg placebo implant)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxandrolone — Absorbable oxandrolone implant (subdermal insertion) Men: 400 mg oxandrolone (two 200 mg oxandrolone implants each) Women: 200 mg oxandrolone (one 200 mg oxandrolone implant)
  Arms: Oxandrolone
Drug: Placebo — Absorbable placebo implant (excipients; subdermal insertion) Men: 400 mg placebo (two 200 mg placebo implants each) Women: 200 mg placebo (one 200 mg placebo implant)
  Arms: Placebo

SUMMARY:
Rehabilitation of knee stability and function after anterior cruciate ligament (ACL) reconstruction is slow and costly. The use of anabolic steroids, such as oxandrolone, may aid in the recovery of muscle mass and strength, as well as functional capacity. Oxandrolone, derived from dihydrotestosterone, has high anabolic activity and low androgenic activity (a 13:1 ratio), making it more effective in promoting weight gain with fewer side effects compared to other steroids. Registered by the FDA and previously by ANVISA (National Health Surveillance Agency (Brazil), it is indicated for cases of post-trauma or post-surgery weight loss. The subdermal use of oxandrolone implants is proposed to release the drug directly into the bloodstream, improving efficacy and reducing issues related to oral administration. This study evaluates the safety and tolerability of the absorbable subdermal oxandrolone implant for 24 weeks versus placebo implant in both men and women as an adjuvant treatment during rehabilitation following anterior cruciate ligament (ACL) surgical reconstruction. The serum and pharmacokinetic profile of the oxandrolone implant will be monitored.

DETAILED DESCRIPTION:
This is a phase II, randomized, double-blind, placebo-controlled, multicenter clinical study designed to evaluate the safety and tolerability profile of the absorbable oxandrolone implant as an adjuvant treatment in rehabilitation following anterior cruciate ligament (ACL) reconstruction surgery. The primary safety outcome will be the incidence of serious adverse events (SAEs) collected through spontaneous reports and/or clinical findings over 24 weeks after randomization (subdermal insertion of the absorbable oxandrolone implant). The exploratory evaluation of the efficacy of the absorbable oxandrolone implant will compare the use of oxandrolone implant with a placebo pellet in the rehabilitation of patients after ACL reconstruction surgery will be based on its effects on muscle mass recovery, muscle strength, and functional capacity.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged between 18 and 45 years old
* Body weight between 50-110 kg for men and 40-90 kg for women
* BMI ≤30
* Complete rupture of the ACL as visualized by pre-operative magnetic resonance imaging
* Pre-operative radiographic examination with normal joint condition
* Having undergone knee arthroscopy surgery for anterior cruciate ligament reconstruction using autologous hamstring tendon graft
* No other associated injuries, such as posterior cruciate ligament (PCL) injury, grade III medial collateral ligament (MCL) injury, or severe concomitant injury in the contralateral knee (LCL)
* Very active, active, or irregularly active classification of type A or B by the International Physical Activity Questionnaire (IPAQ)
* Continuation of meeting all inclusion criteria verified at the Screening Visit (SV/V1).
* Adherence to the rehabilitation protocol, having participated in at least 10 physical therapy sessions since the SV/V1.
* Functional range of motion from 0 to 120º and ability to walk without the aid of crutches.
* Sitting blood pressure in the clinic <180/95 mmHg.
* Hematocrit ≤ 50%.
* ALT less than three times the upper limit of normal.
* Serum creatinine <2 mg/dl.
* Bilirubin < 3.0 mg/dl.
* Albumin <3 g/dl or prealbumin <10 mg/dl.
* PSA ≤ 4.1 ng/ml (men only).

Exclusion Criteria:

* Only for female participants:
* Confirmed or suspected pregnancy
* History of childbirth, miscarriage, or lactation within the past 3 months
* Refusal to use permitted contraceptive methods during the study and for 90 days after study completion, unless surgically sterile or expressly declaring to be at no risk of pregnancy due to abstinence or non-reproductive sexual practices
* Clinical signs of hyperandrogenism
* Polycystic Ovary Syndrome (PCOS)
* Known or suspected breast carcinoma

Only for male participants:

-Known or suspected prostate or male breast carcinoma

For both male and female participants:

* Previous severe injury or history of surgery on the lower limbs
* Knee injury older than 12 months
* Unstable longitudinal meniscal tear
* Meniscus suture during ACL surgical reconstruction
* Use of patellar, quadriceps, or any graft other than hamstring tendon during ACL surgical reconstruction
* Known contraindication to hormone use
* Any condition that worsens with hormonal treatment
* Personal history of deep vein thrombosis (DVT)
* Known coagulopathy
* Known chromosomal disorders
* Hypersensitivity to anabolic androgenic steroids
* Previous failure of oxandrolone treatment
* Use of testosterone (or analogs) and other anabolic androgenic steroids in any pharmaceutical form within the last 3 months
* Pituitary tumor
* Creatinine levels >2 mg/dl or history of chronic kidney disease
* Myocardial infarction within the last 6 months
* Uncontrolled dyslipidemia
* Uncontrolled diabetes
* Patients with chronic obstructive pulmonary disease (COPD) not responsive to bronchodilators
* Any contraindication to undergoing magnetic resonance imaging (MRI)
* Claustrophobia
* Sedentary classification according to the International Physical Activity Questionnaire (IPAQ)
* High-performance athlete
* Known psychiatric diagnosis, including major or persistent depressive disorder, bipolar disorder, anxiety disorders, social phobia, specific phobias, obsessive-compulsive disorder, psychotic disorders, personality disorders, eating disorders, neurocognitive disorders, developmental disorders, or somatoform disorders (somatization or hypochondriasis)
* Presence of urinary disorders
* Known diagnosis of fibromyalgia
* Current smoking
* History of drug abuse
* Participation in other clinical trial protocols within the past 30 days
* Participant who, in the investigator's opinion, presents other conditions or clinical/laboratory abnormalities that make them unsuitable to participate in the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-10-31 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Combination of serious adverse events (SAEs) accumulated within 24 weeks of oxandrolone or placebo pellet insertion and collected through spontaneous reporting and/or clinical findings | From randomization to the end of study on Week 24.
  Proportion of patients who do NOT have SAEs: defined as a combination of death, conditions that threat or present risk to life, conditions needing hospitalization or prolonging the pre-existing hospitalization, conditions causing disability or permanent damage, conditions leading to a congenital anomaly and any other significant medical occurrence that, based on appropriate medical judgment, may harm the participant and/or require medical or surgical intervention to prevent any of the other aforementioned occurrences.

SECONDARY OUTCOMES:
Biochemical Profile | At pre-insertion, 4, 12, and 24 weeks after randomization
  Combination of the number of participants who present laboratory test values of the biochemical profile (safety) outside the reference range and clinically significant for 24 weeks after randomization.
  Laboratory tests (biochemical profile):
  • Men and women: Hematocrit, Platelet count, Serum creatinine, Serum urea, Total bilirubin, Aspartate aminotransferase (AST/TGO), Alanine aminotransferase (ALT/TGP), Alkaline phosphatase (FA), Gamma-glutamyl transferase (GGT), Creatine phosphokinase (CPK).
  • Only in Men: Serum levels of Prostate-Specific Antigen (PSA).
Metabolic Profile | At pre-insertion, 4, 12, and 24 weeks after randomization
  Combination of the number of participants who present laboratory test values of the metabolic profile outside the reference range and clinically significant for 24 weeks after randomization.
  Laboratory tests (metabolic profile):
  • Men and women: Total cholesterol, LDL, HDL, Lipoprotein.
Hormonal Profile | At pre-insertion, 4, 12, and 24 weeks after randomization
  Combination of the number of participants who present laboratory test values of the hormonal profile outside the reference range and clinically significant for 24 weeks after randomization.
  Laboratory tests (hormonal profile):
  • Men: Serum concentration of total and free testosterone, Serum concentration of follicle-stimulating hormone (FSH), Serum concentration of luteinizing hormone (LH), Serum concentration of sex hormone-binding globulin (SHBG).
Hemostasis Parameters | At pre-insertion, 4, 12, and 24 weeks after randomization
  Combination of the number of participants who present laboratory test values of hemostasis parameters outside the reference range and clinically significant for 24 weeks after randomization.
  Laboratory tests (hemostasis parameters):
  • Men and women: D-dimer, SHBG, Free Protein S,
Total serum oxandrolone concentration | Pre-insertion of the oxandrolone implant; various times after the insertion of the oxandrolone implant and 24 hours; 1, 2, 3, 4, 8, 12, 16, 20, and 24 weeks.
  Multiple blood sample will be collected at various times after randomization for those who agree to participate (SUBGROUP; N=20 men and women) and total serum oxandrolone will be determined by liquid chromatography (LC-MS/MS).
Area under the curve (AUC(0 ∞)) | Pre-insertion of the oxandrolone implant and various times after the insertion of the oxandrolone implant: 24 hours; 1, 2, 3, 4, 8, 12, 16, 20, and 24 weeks.
  Multiple blood sample will be collected at various times after randomization for those who agree to participate (SUBGROUP; N=20 men and women) and will be determined by liquid chromatography (LC-MS/MS).
Maximum concentration (Cmax) | Pre-insertion of the oxandrolone implant and various times after the insertion of the oxandrolone implant: 24 hours; 1, 2, 3, 4, 8, 12, 16, 20, and 24 weeks.
  Multiple blood sample will be collected at various times after randomization for those who agree to participate (SUBGROUP; N=20 men and women) and will be determined by liquid chromatography (LC-MS/MS).
Time to reach maximum concentration (tmax) | Pre-insertion of the oxandrolone implant and various times after the insertion of the oxandrolone implant: 24 hours; 1, 2, 3, 4, 8, 12, 16, 20, and 24 weeks.
  Multiple blood sample will be collected at various times after randomization for those who agree to participate (SUBGROUP; N=20 men and women) and will be determined by liquid chromatography (LC-MS/MS).
Half Life (t1/2) | Pre-insertion of the oxandrolone implant and various times after the insertion of the oxandrolone implant: 24 hours; 1, 2, 3, 4, 8, 12, 16, 20, and 24 weeks.
  Multiple blood sample will be collected at various times after randomization for those who agree to participate (SUBGROUP; N=20 men and women) and will be determined by liquid chromatography (LC-MS/MS).

OTHER OUTCOMES:
Changes in body composition | At pre-insertion and 12 and 24 weeks after randomization
  Distribution and percentages of lean mass and fat by bioimpedance
Changes in maximal muscle strength using isometric dynamometry | At pre-insertion, 12 and 24 weeks after randomization
  To assess isometric strength, a Lafayette handheld isometric dynamometer or its national equivalent will be used. The evaluation will be conducted for the knee extensors and flexors. The parameters used in the assessment are defined by the literature: normalization and symmetry index; peak torque (Nm) of the quadriceps; limb symmetry index (LSI).
Changes in the Short Form Health Survey SF-36 Quality of Life Questionnaire | At pre-insertion, 12 and 24 weeks after randomization
  Number of participants with changes in the 36-Item Short Form Health Survey (SF-36). SF-36 is a patient-reported outcome (PRO) measure evaluating a participant's health status. It comprises 36 items covering 8 domains: physical functioning, role physical, role emotional, bodily pain, vitality, social functioning, mental health, and general health. Items are answered on Likert scales of varying lengths. Items from 8 domains contribute to the PCS. The summary scores range from 0 to 100, with higher scores indicating better levels of function and/or better health
Changes in the General Anxiety Disorder Questionnaire (GAD-7) | At pre-insertion, 12 and 24 weeks after randomization
  The GAD-7 is a self-administered questionnaire that assesses generalized anxiety, composed of seven questions covering aspects such as excessive worry, difficulty controlling worry, irritability, muscle tension, fatigue, difficulty relaxing, and sleep problems. Each question is scored from 0 to 3, with a severity score ranging from 0 to 21. Cutoff points are ≥5 for mild anxiety, ≥10 for moderate anxiety, and ≥15 for severe anxiety.
Changes in the Patient Health Questionnaire (PHQ-9) | At pre-insertion, 12 and 24 weeks after randomization
  The PHQ-9 is a self-administered questionnaire focused on depression, consisting of nine questions addressing aspects like diminished interest, depressed mood, fatigue, sleep issues, appetite changes, low self-esteem, difficulty concentrating, slowed movements or agitation, and suicidal thoughts. Each question is scored from 0 to 3, with a severity score from 0 to 27. Severe depression is indicated by a score >16.
Changes in the Patient Acceptable Symptom State (PAS) | At pre-insertion, 12 and 24 weeks after randomization
  The PAS is a method used to assess whether the current symptom state of a patient is acceptable to them, considering their personal perspective of well-being and functionality. It consists of a single standardized question that captures the patient's global satisfaction with their current condition.
Changes in the Knee Society Score (KSS) | At pre-insertion, 12 and 24 weeks after randomization
  The KSS is an assessment used to measure knee function and pain in patients who have undergone orthopedic knee surgeries. It assesses postoperative recovery, quality of life, and treatment effectiveness. The KSS consists of two main components: 1) Functional KSS: Assesses knee function in terms of mobility and the ability to perform daily activities (such as walking, climbing stairs, sitting and standing, etc.); 2) Pain KSS. It integrates the patient's ability to perform common tasks without significant pain or difficulty. The score ranges from 0 to 100, with 100 indicating the best performance (no difficulties in functional activities) and 0 indicating the worst (total inability to perform these activities).
Changes in the Y Balance Test | 12 and 24 weeks after randomization
  The Y Balance Test is a functional assessment used to measure mobility, muscle strength, and trunk and lower limb stability. It is used to identify muscle imbalances, strength deficiencies, and injury risks in individuals recovering from injuries. The final test score is the distance reached in each direction, expressed as a percentage of leg length (adjusting the results based on body size). Comparisons are made between limbs (right leg vs. left leg) to check for symmetry and identify possible deficiencies or imbalances. The patient must achieve less than 4cm of anterior reach difference between legs.
Changes in the Lysholm Knee Scoring Scale | At pre-insertion, 12 and 24 weeks after randomization
  The Lysholm Knee Scoring Scale provides a quantification of knee function, allowing comparison of a patient's progress over time. It consists of 8 items. These items are divided into two categories: (1) Symptoms, which evaluate pain, locking, and instability; and (2) Function, which assesses the ability to climb stairs, run, perform daily activities, and squat. The participant responds to each item, which is scored according to the severity or frequency of the symptoms. The total score ranges from 0 to 100 points, with 100 representing the best possible outcome (indicating ideal knee function) and 0 representing the worst outcome (indicating severe dysfunction or disability of the knee).

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Tauchmann, MD, Principal Investigator — Hospital do Rocio
Locations (2):
- Brazil (2):
  - Santa Casa de Santos, Santos, São Paulo
  - Science Valley Research Institute, São Paulo, Sao Paulo, São Paulo, São Paulo

REFERENCES:
- [Background] Bakowski P, Bakowska-Zywicka K, Piontek T. Clinical practice and postoperative rehabilitation after knee arthroscopy vary according to surgeons' expertise: a survey among polish arthroscopy society members. BMC Musculoskelet Disord. 2020 Sep 23;21(1):626. doi: 10.1186/s12891-020-03649-9. PMID 32967668